CLINICAL TRIAL: NCT00061997
Title: A Phase I Study Of The Safety Of Myo-Inositol As A Chemopreventive Agent
Brief Title: Inositol in Preventing Lung Cancer in Patients With Bronchial Epithelial Dysplasia Who Are Current or Former Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Prevention
Other Study IDs: CDR0000302633; BCCA-U98-0411; BCCA-C02-0298
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2005-11

CONDITIONS: Lung Cancer; Precancerous Condition
Keywords: non-small cell lung cancer; small cell lung cancer; precancerous condition
MeSH Terms: conditions — Lung Neoplasms; Precancerous Conditions; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Inositol

INTERVENTIONS:
Dietary Supplement: inositol

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. Inositol may be effective in preventing the development of lung cancer in patients with bronchial epithelial dysplasia.

PURPOSE: This phase I trial is studying the side effects and best dose of inositol in preventing lung cancer in current or former smokers with bronchial epithelial dysplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of inositol for the prevention of lung cancer in patients with bronchial epithelial dysplasia who are current or former smokers.
* Determine the potential efficacy of this drug in regression of existing dysplastic lesions or prevention of appearance of new dysplastic lesions in these patients.
* Determine whether intake of this drug can facilitate smoking cessation in patients who are current smokers.

OUTLINE: This is a dose-escalation study.

Patients receive oral inositol twice daily. Treatment continues for 1 or 3 months in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-12 patients receive escalating doses of inositol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 12 patients experience dose-limiting toxicity.

Once the MTD is determined, 10 patients are treated with inositol twice daily at the MTD for 3 months in the absence of disease progression or unacceptable toxicity.

Patients are followed at 1 month.

PROJECTED ACCRUAL: A total of 3-28 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of persistent bronchial dysplasia despite regular twice-daily treatment with inhaled budesonide for 6 or 12 months on protocol BCCA-CIC-98-37
* Current or former smokers who have smoked at least 30 pack years
* Sputum cells showing AIC atypia by computer-assisted image analysis
* At least 2 abnormal sites on fluorescence bronchoscopy (red/green ratio at least 0.45) suspicious for bronchial dysplasia

  * At least 1 site confirmed by bronchial biopsy
  * Solitary dysplastic lesion allowed provided the diameter is greater than 1.5 mm
* No invasive cancer on bronchoscopy or abnormal low-dose spiral CT scan suspicious for lung cancer

PATIENT CHARACTERISTICS:

Age

* 40 to 74

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Hematologic function normal
* No bleeding disorder

Hepatic

* Liver function normal
* Liver enzymes no greater than upper limit of normal

Renal

* Renal function normal

Cardiovascular

* No unstable angina
* No congestive heart failure

Pulmonary

* No acute or chronic respiratory failure
* No acute bronchitis or pneumonia within the past month

Other

* Fasting glucose less than 144 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing to have a bronchoscopy
* No schizophrenia
* No bipolar disorder
* No diabetes
* No known reaction to topical xylocaine
* No other medical condition that would jeopardize patient safety during study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

Surgery

* No prior surgery for lung cancer

Other

* No concurrent lithium

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-05

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lam, MD, Study Chair — British Columbia Cancer Agency
Locations (1):
- British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia, Canada